CLINICAL TRIAL: NCT05387538
Title: One-layer Versus Two-layer Duct-to-mucosa Pancreaticojejunostomy After Pancreaticoduodenectomy : Randomized Comparative Prospective Study .
Brief Title: One-layer Versus Two-layer Duct-to-mucosa Pancreaticojejunostomy After Pancreaticoduodenectomy .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr. Hamada, assistant lecturer at general surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HF2022
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Fistula
Keywords: Pancreaticojejunostomy; Duct-to-mucosa
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Intervention Model Description: patients will be randomized into two groups according to the surgical procedure performed as follows group (A )had pts who will undergo One-layer Duct-to-mucosa Pancreaticojejunostomy group(B) had pts who will undergo Two-layer Duct-to-mucosa Pancreaticojejunostomy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-layer Duct-to-mucosa Pancreaticojejunostomy (Experimental): pancreatic anastomosis to jejunum will be performed in one layer suturing the pancreatic duct to the mucosa of jejunum.
  Interventions: Procedure: One-layer Duct-to-mucosa Pancreaticojejunostomy
- Two-layer Duct-to-mucosa Pancreaticojejunostomy (Experimental): pancreatic anastomosis to jejunum will be performed in two layer. The first layer will be suturing the pancreatic capsule to the seromuscular layer of jejunum and the 2nd layer will be suturing the pancreatic duct to the mucosa of jejunum.
  Interventions: Procedure: Two-layer Duct-to-mucosa Pancreaticojejunostomy

INTERVENTIONS:
Procedure: One-layer Duct-to-mucosa Pancreaticojejunostomy — To create the anterior suturing layers, double needles with a 4/0 or 3/0 Prolene line will be used; one side of the needles will be inserted from the anterior inner side of the pancreatic duct and out through the ventral parenchyma of the pancreatic stump to the anterior surface of the pancreas about 3 cm from the cut edge. The other side of the needles will be started from the inner side of the jejunum lumen, then pushed through the subserosa and seromuscular region, and out from the posterior surface of the bowel but its done after completion of the posterior layer. The posterior suturing layer will be treated in the same manner. An internal pancreatic duct stent will be used
  Arms: One-layer Duct-to-mucosa Pancreaticojejunostomy
Procedure: Two-layer Duct-to-mucosa Pancreaticojejunostomy — The same double needle and 4/0 or 3/0Prolene line will be used. First, the region approximately 1.0 cm from the cutting edge of the pancreatic remnant will be freed; then, the posterior surface of the pancreatic remnant will be sutured to the seromuscular layer of the jejunum using the interrupted suturing method. The jejunum will be brought closer to the stump of the pancreas, and a hole of similar diameter to the main pancreatic duct will be made on the jejunum near the entrance of the main pancreatic duct. The posterior wall of the jejunum near the hole will be sutured to the posterior wall of the pancreatic duct using the interrupted suturing method with Prolene line, and a suitable internal pancreatic duct stent will used . The interior side of the jejunum and pancreas will be sutured using the same method. Then, the anterior surface of the pancreatic remnant and the seromuscular layer of the jejunum will be tightly sutured using the interrupted method.
  Arms: Two-layer Duct-to-mucosa Pancreaticojejunostomy

SUMMARY:
Postoperative pancreatic fistula (POPF) is one of the most frequent and ominous complications after PD, and its occurrence reportedly ranges from 2-40 %. Severe POPF prolongs hospital stay and requires the use of specific treatments, such as the use of antibiotics, nutritional support, endoscopy, interventional radiology, and/or reoperation, etc.. Several anastomotic surgical techniques have been developed to reduce the incidence of pancreatic fistula in recent decades, including the duct-to-mucosa method, pancreaticogastrostomy, Peng's binding method, and the "end-to-end" or "end-to-side" invaginated method. Among these techniques, the conventional duct-to-mucosa method remains the most popular anastomosis due to its advantages.

The size of the pancreatic remnant is not limited; moreover, the jejunal lumen and pancreatic remnant lead to easier anastomosis . Compared with two-layer duct-to-mucosa anastomosis, the novel one-layer duct-to-mucosa PJ anastomosis method has been reported to be efficient at reducing POPF occurrence. However, the two cited retrospective studies might lead to selection bias. Because this evidence is insufficient, we will conduct a randomized controlled trial to verify the superiority of one-layer duct-to-mucosa PJ anastomosis after PD over the two-layer technique.

DETAILED DESCRIPTION:
To date, pancreaticoduodenectomy (PD) has been regarded as the only potentially curative treatment for pancreatic head and periampullary tumors, including tumors in the ampullary region, distal biliary duct, and periampullary duodenum .

A retrospective study in which 1000 cases were recruited over the past three decades showed that PD has become an effective treatment to reduce hospital mortality. Mortality has been reduced to less than 5 %, but the morbidity remains at 30-50 % .

Postoperative pancreatic fistula (POPF) is one of the most frequent and ominous complications after PD, and its occurrence reportedly ranges from 2-40 %. Severe POPF prolongs hospital stay and requires the use of specific treatments, such as the use of antibiotics, nutritional support, endoscopy, interventional radiology, and/or reoperation, etc.

POPF risk is increased by many factors including pancreatic texture, main pancreatic duct diameter, and pancreaticojejunal (PJ) anastomotic technique .Among these factors, only anastomotic technique can be improved. According to the International Study Group of Pancreatic Surgery (ISGPS) definition, POPF exists if the drainage of any measurable volume of fluid containing amylase exceeds three times the normal serum value on or after postoperative day (POD) 3.

Several anastomotic surgical techniques have been developed to reduce the incidence of pancreatic fistula in recent decades, including the duct-to-mucosa method, pancreaticogastrostomy, Peng's binding method, and the "end-to-end" or "end-to-side" invaginated method. Among these techniques, the conventional duct-to-mucosa method remains the most popular anastomosis due to its advantages.

The size of the pancreatic remnant is not limited; moreover, the jejunal lumen and pancreatic remnant lead to easier anastomosis .Compared with two-layer duct-to-mucosa anastomosis, the novel one-layer duct-to-mucosa PJ anastomosis method has been reported to be efficient at reducing POPF occurrence . However, the two cited retrospective studies might lead to selection bias. Because this evidence is insufficient, we will conduct a randomized controlled trial to verify the superiority of one-layer duct-to-mucosa PJ anastomosis after PD over the two-layer technique.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, aged 18 to 65. Patients scheduled to undergo pancreaticoduodenectomy.

Exclusion Criteria:; Patients who had a previous pancreatic operation; Patients with an immunodeficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pancreatic fistula(POPF) rate | 30 days
  drainage of any measurable volume of fluid with an amylase content >3 times the upper normal serum value on or after postoperative day 3.

SECONDARY OUTCOMES:
Duration of postoperative hospital stay | 30 days
  Time from day of operation to day of discharge
anastomosis time | 1 hour
  anastomosis time was calculated from beginning to the end of pancreaticojejunostomy

CONTACTS AND LOCATIONS:
Overall Officials: Abd El-moniem I.M El-khateeb, professor, Study Chair — Faculty of medicine_Assuit university_Assuit_ Egypt

IPD SHARING:
Plan to Share IPD: Undecided